CLINICAL TRIAL: NCT03164395
Title: The Efficacy of Single Coil Defibrillation Leads for Internal Cardioversion of Persistent Atrial Fibrillation
Brief Title: The Efficacy of Single Coil Defibrillation Leads for Internal Cardioversion of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Samy C Elayi, MD, Assistant Professor, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-0536
Record Dates: First submitted 2017-05-21; First posted 2017-05-23 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; implantable cardiac defibrillator; cardioversion
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in block fashion to either internal or external cardioversion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal Cardioversion (Experimental): Patients randomized to external cardioversion will undergo external synchronized cardioversion per institutional protocol.
  Interventions: Procedure: Internal Cardioversion
- External Cardioversion (Active Comparator): Patients randomized to internal cardioversion will have a maximum energy shock delivered from the device between the RV coil and can. If cardioversion is not successful they will then undergo external cardioversion per institutional protocol.
  Interventions: Procedure: External Cardioversion

INTERVENTIONS:
Procedure: Internal Cardioversion — Internal Cardioversion with device maximum output shock from RV coil to Can versus external cardioversion per institutional protocol
  Arms: Internal Cardioversion
Procedure: External Cardioversion — External Cardioversion per institutional protocol
  Arms: External Cardioversion

SUMMARY:
This study seeks to determine the efficacy of single coil defibrillation leads for cardioversion of persistent atrial fibrillation.

DETAILED DESCRIPTION:
This study seeks to compare the efficacy of single coil defibrillation leads for the internal cardioversion of atrial fibrillation as compared with cardioversion by external defibrillation pads. It is known that dual coil leads are effective for atrial cardioversion, but the presence of the SVC defibrillation coil allows for selection of shock vector that more reliably incorporates the majority of atrial tissue compared to a single right ventricular lead. For a variety of reasons single coil defibrillation leads are now implanted in the majority of patients requiring placement of implantable cardiac defibrillators, and many of these patient's will later develop atrial fibrillation and potentially require cardioversion. Currently, there is no clear consensus on how to approach cardioversion in these patient's and both external and internal methods are used. Internal cardioversion may be ineffective exposing patient's unnecessarily to repeated shocks and battery depletion. External cardioversion may carry a small risk of damaged to the CIED.

The investigator's goal is to identify patient's referred for cardioversion for atrial fibrillation who also have an implanted cardiac defibrillator with a single coil defibrillation lead and randomize them to either external or internal cardioversion.

ELIGIBILITY:
Inclusion Criteria:

* greater than 18 years of age
* persistent atrial fibrillation and have been recommended by your primary cardiologist to undergo cardioversion
* have an implantable cardiac defibrillator

Exclusion Criteria:

* over the age of 99
* pregnant
* prisoner

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
Acute Conversion of Atrial Fibrillation to Sinus Rhythm | Immediate
  Does the patient return for at least one beat to sinus rhythm following the administration of a shock

CONTACTS AND LOCATIONS:
Overall Officials: Samy C Elayi, MD, Study Chair — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No